CLINICAL TRIAL: NCT02791152
Title: SingHEART: Effects of Physical Activity, Ambulatory Blood Pressure and Calcium Score on Cardiovascular Health in Normal People
Brief Title: Effects of Physical Activity, Ambulatory Blood Pressure and Calcium Score on Cardiovascular Health in Normal People
Acronym: SingHEART
Status: Recruiting | Type: Observational
Sponsor: National Heart Centre Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2015/2601
Record Dates: First submitted 2016-05-31; First posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2015-09

CONDITIONS: Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A prospective cohort of relatively healthy individuals, using comprehensive clinical information, advanced imaging (including cardiac MRI), cardiovascular exercise physiology, metabolomics and genetic analysis. These findings will be correlated with adverse clinical outcomes including death, stroke and myocardial infarction. In selected cases, follow-up imaging and biomarker samples will also be obtained. These studies will enable us to begin to address a critical gap in our knowledge as to how best to interpret the very large amount of cardiovascular tests done in Singapore and how to better to predict outcomes and manage healthcare costs in our local populations

DETAILED DESCRIPTION:
SingHEART sub-study will collect the following data types or perform the following investigations:

1. Demographic and clinical characteristics data.
2. Basic blood investigations. Basic blood investigations include: FBC, CRP, renal panel, random glucose, LFT, fasting lipids, ESR, CRP,
3. Perform a single baseline cardiac MRI (already consented and obtained as part of the primary study).
4. ECG
5. Calcium score
6. Biobanking (whole blood, plasma and serum, already performed as part of the primary study)
7. Exercise and physical activity tracker over two 1-week periods
8. Ambulatory BP monitoring over two 24-48H periods

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 21-69 years

Exclusion Criteria:

1. Previous myocardial infarction (MI). This will include ST-elevation MI (STEMI) and non-ST-elevation MI (NSTEMI)
2. Known coronary artery disease - prior coronary revascularization
3. Known documented peripheral arterial disease
4. Previous stroke

   a. Stroke is defined as new focal neurological deficit persisting more than 24hours21.
5. More than ongoing use of 2 or more anti-hypertensive agents
6. Prior history of cancer (excludes pre-cancerous lesions)
7. Expected life expectancy less than 1 year
8. Known definite diabetes mellitus or on treatment for diabetes mellitus
9. Known autoimmune disease or genetic disease
10. Known endocrine disease on treatment
11. Psychiatric illness
12. Asthma or chronic lung disease requiring long term medications or oxygen
13. Chronic infective disease, including tuberculosis, hepatitis B and C; and HIV
14. Inability to comply with study protocol
15. Any other acute or chronic medical or physical condition deemed by the investigator to affect study outcomes

Ages: 21 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers age between 21 to 69 years old, Singapore citizens
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2015-10; Primary Completion 2036-12 (Estimated); Study Completion 2036-12 (Estimated)

PRIMARY OUTCOMES:
First cardiovascular event | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Yeo Khung Keong, MBBS, Principal Investigator — National Heart Centre Singapore
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bylstra Y, Lim WK, Teo JX, Menezes M, Hodgson J, Yap F, Chambers JC, Yeo KK, Tan P, Amor DJ, Jamuar SS. Unexpected genotypes associated with severe paediatric conditions identified in a healthy population cohort. Eur J Hum Genet. 2026 Jan 10. doi: 10.1038/s41431-025-02009-2. Online ahead of print. PMID 41520097
- [Derived] Bylstra Y, Lim WK, Kam S, Tham KW, Wu RR, Teo JX, Davila S, Kuan JL, Chan SH, Bertin N, Yang CX, Rozen S, Teh BT, Yeo KK, Cook SA, Jamuar SS, Ginsburg GS, Orlando LA, Tan P. Family history assessment significantly enhances delivery of precision medicine in the genomics era. Genome Med. 2021 Jan 7;13(1):3. doi: 10.1186/s13073-020-00819-1. PMID 33413596